CLINICAL TRIAL: NCT07074015
Title: IntelliWell: An AI-Assisted Microwell Platform for Label-Free Localization of Ultra-Rare Sperm in Non-Obstructive Azoospermia Micro-TESE Specimens
Brief Title: IntelliWell: An AI-Assisted Imaging Platform for Detection and Location of Ultra-Rare Testicular Sperm in Surgical Specimens
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Martin Kathrins, M.D., Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025p001209
Record Dates: First submitted 2025-05-19; First posted 2025-07-20 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Infertility; Azoospermia
Keywords: infertility; azoospermia; micro-TESE
MeSH Terms: conditions — Infertility; Azoospermia | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- IntelliWell Arm (Experimental)
  Interventions: Device: Use of IntelliWell to identify and localize sperm for ICSI

INTERVENTIONS:
Device: Use of IntelliWell to identify and localize sperm for ICSI — The experimental arm will have surgically extracted testicular sperm processed with IntelliWell. If identified and confirmed by embryology, cryopreservation of sperm will occur. On day of ICSI, thaw of testicular sperm will occur and be processed by IntelliWell for identification and localization for use in ICSI.

SUMMARY:
This study will help determine whether an AI-assisted microwell platform (IntelliWell) can identify rare sperm cells in testicular samples found to not have sperm by conventional analysis. Instead of discarding testicular tissue which was found to be non-sperm bearing by conventional analysis the testicular tissue will be processed using IntelliWell and, if sperm is found and verified by embryologists, it may be used for intracytoplasmic sperm injection (ICSI).

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects presenting to Brigham and Women's or Faulkner urology clinic with infertility with clinical non-obstructive azoospermia (clinical diagnosis based on two semen analyses, physical examination, and hormonal testing).
2. Male subjects undergoing micro-surgical testicular sperm extraction surgery at Brigham and Women's Hospital.
3. Surgically extracted sperm which are not found to have clinically usable quantities of sperm after standard of care manual processing for which samples would otherwise be discarded and the procedure deemed unsuccessful.

Exclusion Criteria:

1. Female subject (with whom male subjects intends to conceive with surgically extracted sperm) cannot or will not provide her informed consent for study participation. She will undergo ICSI at BWH with BWH embryology.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-02-15 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Sperm detection rate by IntelliWell (sperm/min) | Date of surgery and date of ICSI
Sperm retrieval success rate | Date of surgery and date of ICSI
  Defined as at least one ICSI-grade sperm retrieved from IntelliWell

SECONDARY OUTCOMES:
Total number of sperm detected in IntelliWell in fresh sample | Date of surgery
Total number of sperm detected by IntelliWell in test-thaw samples | Day of surgery
Total number of sperm detected by IntelliWell on day of ICSI | Date of ICSI
Time to first sperm detection and time to 10 sperm | Date of surgery and date of ICSI
Number of IntelliWell-identified sperm verified by embryology | Date of surgery and date of ICSI
Number of sperm retrieved and approved for ICSI | Date of ICSI
Total IntelliWell search time | Date of surgery and date of ICSI

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kathrins M, Abhyankar N, Shoshany O, Liebermann J, Uhler M, Prins G, Niederberger C. Post-thaw recovery of rare or very low concentrations of cryopreserved human sperm. Fertil Steril. 2017 Jun;107(6):1300-1304. doi: 10.1016/j.fertnstert.2017.04.016. Epub 2017 May 5. PMID 28483505
- [Background] Bernie AM, Mata DA, Ramasamy R, Schlegel PN. Comparison of microdissection testicular sperm extraction, conventional testicular sperm extraction, and testicular sperm aspiration for nonobstructive azoospermia: a systematic review and meta-analysis. Fertil Steril. 2015 Nov;104(5):1099-103.e1-3. doi: 10.1016/j.fertnstert.2015.07.1136. Epub 2015 Aug 8. PMID 26263080
- [Background] Berger AJ, Raup V, Abou Ghayda R, Lanes A, Kathrins M. Inability to obtain sperm for fresh IVF cycles: analysis and incidence of outcomes using a database from the United States. Fertil Res Pract. 2020 Aug 11;6:14. doi: 10.1186/s40738-020-00082-3. eCollection 2020. PMID 32793376